CLINICAL TRIAL: NCT00064974
Title: A Multicenter, Single-Arm, Open-Label Study of the Efficacy and Safety of CC-5013 Monotherapy in Subjects With Myelodysplastic Syndromes
Brief Title: Efficacy and Safety Study of CC-5013 Monotherapy in Subjects With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Celgene (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MDS-002; NCT00077506 (obsolete NCT alias)
Record Dates: First submitted 2003-07-16; First posted 2003-07-17 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS; CC-5013; Revlimid; Celgene
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CC-5013 (Experimental): CC-5013 10 mg (two 5 mg capsules) daily on days 1-28 every 28 days (28 day cycles)
  Interventions: Drug: CC-5013

INTERVENTIONS:
Drug: CC-5013 — CC-5013 10 mg (two 5 mg capsules) daily on days 1-28 every 28 days (28 day cycles)
  Other Names: lenalidomide

SUMMARY:
This study is a multi-center, single-arm, open-label study of oral CC-5013 monotherapy administered at a dose of 10 mg daily on Days 1-21 every 28 days (28-day cycles) to red blood cell (RBC) transfusion-dependent subjects with low- or intermediate-1-risk MDS who do not have a del (5q31-33) cytogenetic abnormality. Screening procedures will take place within 28 days of first day of study drug treatment. Subjects will receive study drug (CC-5013) in 28-day cycles for up to 6 cycles, or until bone marrow disease progression or progression/relapse following erythroid hematologic improvement (Appendix I) is documented. Study visits will occur every cycle (every 28 days) and laboratory monitoring to assess hematological parameters will occur every 14 days. Safety and efficacy assessments to be performed during the study are outlined in the Schedule of Study Assessments.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form.
* Age ≥ 18 years at the time of signing the informed consent form.
* Must be able to adhere to the study visit schedule and other protocol requirements.
* Diagnosis of low - or intermediate-1-risk IPSS (Appendix III) MDS without an abnormality of chromosome 5 involving a deletion between bands q31 and q33.
* Red blood cell (RBC) transfusion-dependent anemia defined as having received ≥ to 2 units of RBCs within 8 weeks of the first day of study drug treatment.
* Eastern Cooperative Oncology Group (ECOG) (Appendix IV) performance status score of 0, 1, or 2.
* Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test within 7 days of starting study drug.
* Sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on study drug.
* WCBP must agree to have pregnancy tests every 4 weeks while on study drug.

Exclusion Criteria:

* Pregnant or lactating females.
* Prior therapy with lenalidomide.
* An abnormality of chromosome 5 involving a deletion between bands q31 and q33.
* Lab Abnormality: Absolute neutrophil count (ANC) <500 cells/mm3 (0.5 x 109/L)
* Lab Abnormality: Platelet count <50,000/mm3 (50 x 109/L)
* Lab Abnormality: Serum creatinine >2.5 mg/dL (221 mmol/L)
* Lab Abnormality: Serum glutamic oxaloacetic transaminase/Aspartate transaminase (SGOT/AST) or Serum glutamic pyruvic transaminase/Alanine transaminase (SGPT/ALT) >3.0 x upper limit of normal (ULN)
* Lab Abnormality: Serum total bilirubin >2.0 mg/dL (34 mmol/L)
* Prior ≥ grade 3 National Cancer Institute (NCI) Common Toxicity Criteria (CTC) (Appendix VI) allergic reaction/hypersensitivity to thalidomide.
* Prior ≥ grade 3 NCI CTC (Appendix VI) rash or any desquamation (blistering) while taking thalidomide.
* Clinically significant anemia due to factors such as iron, B12 or folate deficiencies, autoimmune or hereditary hemolysis or gastrointestinal bleeding
* If a marrow aspirate is not evaluable for storage iron, transferrin saturation must be > 20 % and serum ferritin not less than 50 ng/mL.
* Use of hematopoietic growth factors within 7 days of the first day of study drug treatment.
* Chronic use (>2 weeks) of greater than physiologic doses of a corticosteroid agent (dose equivalent to >10 mg/day of prednisone) within 28 days of the first day of study drug treatment.
* Use of experimental or standard drugs (i.e. chemotherapeutic, immunosuppressive, and cytoprotective agents) for the treatment of MDS within 28 days of the first day of study drug treatment.
* Prior history of malignancy other than MDS (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast) unless the subject has been free of disease for greater than or equal to 3 years.
* Use of any other experimental therapy within 28 days of the first day of study drug treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2003-06; Primary Completion 2007-01 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
RBC Transfusion Independence

SECONDARY OUTCOMES:
≥ 50% decrease in RBC transfusion requirement
Platelet Response
  Platelet Response
Neutrophil Response
  Neutrophil Response
Bone marrow Response
  Bone marrow Response
Duration of Response
  Duration of Response
Hemoglobin concentration
  Change of hemoglobin concentration from baseline
Number of Participants with Adverse Event
  Number of Participants with Adverse Event

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knight, MD, Study Director — Celgene Corporation
Locations (119):
- United States (38):
  - Arizona Cancer Center, Scottsdale, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Alta Bates Cancer Center, Berkeley, California
  - Desert Hematology Oncology Medical Group, Inc., Rancho Mirage, California
  - Stanford University Medical Center, Stanford, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Cancer & Blood Disease Center, Lecanto, Florida
  - University of Miami- Sylvester Comp Cancer Center, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Northwest Georgia Oncology - Wellstar Cancer Research, Marietta, Georgia
  - Rush Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Midwest Cancer Research Group, Skokie, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University School of Medicine, Detroit, Michigan
  - St. Luke's Oncology and Hematology Associates, Duluth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - St. Vincents Comprehensive Cancer Center, New York, New York
  - New York Hospital- Cornell, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mt. Sinai Medical Center, New York, New York
  - University of Rochester-James P. Wilmot Cancer Center, Rochester, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Kaiser Permanente Northwest Region, Portland, Oregon
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (9):
  - Royal Adelaide Hospital - SA Pathology Haematology, Adelaide, South Australia
  - Princess Alexandra Hospital - Haematology, Brisbane
  - Royal Prince Alfred Hospital - Institute of Haematology, Camperdown
  - Peter McCallum Cancer Institute - Directorate of Cancer Medecine, East Melbourne
  - Frankston Hospital-peninsula Health - Oncology Day Unit, Frankston
  - The Alfred Hospital - malignant haematology & stem cell transplantation, Melbourne
  - Calvary Mater Newcastle - Haematology, Waratah
  - Border Medical Oncology, Wodonga
  - Wollongong Hospital - Haematology, Wollongong
- Belgium (3):
  - UZ Gent - Hematology, Ghent
  - University Hospital Leuven - Hematology, Leuven
  - Cliniques Universitaires ULC de Mont-Godinne - Hematology, Yvoir
- Czechia (2):
  - Fakultní nemocnice Hradec Králové - Hematology, Hradec Králové
  - Charles university Hospital - Internal Medicine, Prague
- Denmark (4):
  - Aalborg Sygemus - Haematology, Aalborg
  - Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense
  - Vejle Hospital - Hematology, Vejle
- France (13):
  - CHU Angers - Service des maladies du sang, Angers
  - Centre Hospitalier de la côte basque - Hematologie, Bayonne
  - Centre Hospitalier Départemental Vendée - Onco-hematologie, La Roche-sur-Yon
  - CHRU de Lille - Service des maladies du sang, Lille
  - Institut Paoli Calmette - Hematology 1, Marseille
  - CHU Hôtel-Dieu - Hematologie, Nantes
  - Hôpital Saint Louis - Immuno-hematologie, Paris
  - CHU Saint Antoine - Service des maladies du sang, Paris
  - CHRU - Hôpital du Haut Lévêque - Centre François Magendie, Pessac
  - Centre Hospitalier Lyon sud - Hematologie, Pierre-Bénite
  - CHRU Hôpital Purpan - Hematologie, Toulouse
  - Hôpital Bretonneau - Hématologie & Thérapie cellulaire, Tours
  - CHU Nancy - Hematologie, Vandœuvre-lès-Nancy
- Germany (8):
  - Universitätsklinikum Essen, Klinik für Hämatologie, Essen
  - Universitätsklinikum Heidelberg - Medizinische Klinik und Poliklinik V, Heidelberg
  - Universitätsklinikum Jena - Klinik fur Innere Medizin II-Hamatologie/Onkologie, Jena
  - Universitätsklinikum Leipzig - Medizinische Klinik und Poliklinik II, Leipzig
  - Universitätsklinikum Münster - Medizinische Klinik und Poliklinik A, Münster
  - Universitätsklinikum Tübingen - Medizinische Klinik und Poliklinik - Abteilung II, Tübingen
  - Universitätsklinikum Ulm - Klinik fur Innere Medizin III, Ulm
  - Universitätsklinikum Würzburg - Medizinische Klinik und Poliklinik II, Würzburg
- University of Athens - Alexandra Hospital; Clinical Therapeutics, Athens, Greece
- Italy (9):
  - Università degli Studi di Bologna - Policlinico S. Orsola - Hematology, Bologna
  - AO Universitaria San Martino - hematooncology, Genova
  - Fondazione "G. Pascale" - Hematology, Napoli
  - Ospedale San Luigi AO Luigi Gonzaga - Hematology, Orbassano
  - Universita degli Studi di Padova - Clinical & Experimental Medicine, Padua
  - Ospedale Guglielmo da Saliceto - hematooncology, Piacenza
  - Unità di Ematologia Arcispedale S. Maria Nuova - Haematology, Reggio Emilia
  - Policlinico Umberto I, Università "La Sapienza" di Roma - Hematology, Roma
  - A.O.U. San Giovanni Battista - Hematology, Torino
- Netherlands (3):
  - VUMC - Hematology, Amsterdam
  - Erasmus Medical Center - Hematology, Rotterdam
  - University Medical Center - Hematology, Utrecht
- Russia (4):
  - Medical Sciences - Hematology & BMT, Moscow
  - Moscow State Medical Institution Municipal Clinical Hospital n.a. S.P. Botkin - Hematology, Moscow
  - Russian Research Institute of Hematology and Blood Transfusion - Hematology, Saint Petersburg
  - State Higher Educational Institution St. Petersburg State Medical University - Onco-hematology, Saint Petersburg
- Spain (8):
  - Hospital Germans Trias i Pujol - Hematology, Badalona
  - Hospital Clinic i Provincial de Barcelona - Hematology, Barcelona
  - Hospital de Donostia - Hematology, Guipúzcoa
  - Hospital de La Princesa - Hematology, Madrid
  - Hospital 12 de Octubre - Hematology, Madrid
  - Hospital de Salamanca - Hematology, Salamanca
  - Hospital Universitario Marqués de Valdecilla - Hematology, Santander
  - Hospital La Fe - Hematology, Valencia
- Sweden (4):
  - Sahlgrenska Hospital, University of Goteborg - Hematology, Gothenburg
  - Karolinska University Hospital Huddinge - Center of hematology, Stockholm
  - Karolinska University Hospital Solna- medicine, Stockholm
  - Overlakare Medocomcentrum - Hematology, Uppsala
- Switzerland (3):
  - Inselspital, Institut für Medizinische Onkologie, Bern
  - Hôpitaux Universitaire de Genève - Oncologie, Geneva
  - Klinik und Poliklinik für Onkologie - UniversitätsSpital Zürich, Zurich
- United Kingdom (10):
  - Royal Bournemouth Hospital - Haematology, Bournemouth
  - St James's University Hospital - Haematology, Leeds
  - St Bartholomew's Hospital - Medical Oncology, London
  - King's College Hospital - Haematology Clinical Trials, London
  - Freeman Hospital - Northern Centre for Cancer Care, Newcastle upon Tyne
  - Nottingham City Hospital - Centre for Clinical Haematology, Nottingham
  - Derriford Hospital - Haematology, Plymouth
  - Royal hallamshire Hospital - Haematology, Sheffield
  - Royal Marsden NHS Foundation Trust - Haematology, Surrey
  - Royal Wolverhampton hospitals trust - Research and development, Wolverhampton

REFERENCES:
- [Derived] Raza A, Reeves JA, Feldman EJ, Dewald GW, Bennett JM, Deeg HJ, Dreisbach L, Schiffer CA, Stone RM, Greenberg PL, Curtin PT, Klimek VM, Shammo JM, Thomas D, Knight RD, Schmidt M, Wride K, Zeldis JB, List AF. Phase 2 study of lenalidomide in transfusion-dependent, low-risk, and intermediate-1 risk myelodysplastic syndromes with karyotypes other than deletion 5q. Blood. 2008 Jan 1;111(1):86-93. doi: 10.1182/blood-2007-01-068833. Epub 2007 Sep 24. PMID 17893227